CLINICAL TRIAL: NCT04836975
Title: A Multicenter Retrospective Observational Study to Reveal the Patterns of Presentation, Management and Outcome of Patients With Small Cell Lung Cancer (SCLC) and Stage III Non-Small Cell Lung Cancer (NSCLC) in Saudi Arabia
Brief Title: Reveal the Patterns of Presentation, Management and Outcome of Patients With SCLC and Stage III NSCLC in Saudi Arabia:
Acronym: REVEAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4191R00036
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: Small Cell Lung Cancer (SCLC); Stage III Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCLC: Patient Diagnosed with Small Cell Lung Cancer- (extensive or limited)
- NSCLC: Patient diagnosed with primary stage III Non-Small cell lung Cancer

SUMMARY:
A retrospective, multi-centre, observational study to describe the treatment patterns, the demographic, clinical outcomes, treatment effectiveness, and healthcare resource utilization (HCRU) for patients diagnosed with primary Small Cell Lung Cancer SCLC (Extensive stage & Limited Stage)and stage III NSCLC in a real-world setting.

DETAILED DESCRIPTION:
A retrospective, multi-centre, observational study to describe the treatment patterns, the demographic, clinical outcomes, treatment effectiveness, and healthcare resource utilization (HCRU) for patients diagnosed with primary Small Cell Lung Cancer SCLC (Extensive stage & Limited Stage)and stage III NSCLC in a real-world setting

Cohort of patients diagnosed with primary SCLC (limited or extensive stage) or stage III NSCLC, aims to characterize the treatment patterns from the index date (defined as the date of initial diagnosis of locally advanced stage III NSCLC and SCLC) to the end of follow-up (defined as the earliest of death, last available medical record or end of the observation period "defined as the date of data abstraction") including the type of treatment received, duration of each treatment regimen, and reasons for stopping treatment regimen.

The study population will be identified by participating physicians involved in the diagnosis, treatment and management of these patients through the review of established patient medical records. Eligible patients (both alive and deceased) will have their data anonymously abstracted from their medical records into a centrally designed electronic case report form (eCRF).

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult male or female (≥18 years old or according to the age of majority as defined by local regulations).

  2. First-ever diagnosis of lung cancer (absence of previous diagnosis of lung cancer, including SCLC and NSCLC) in the patient's medical records.

  3. Patients either diagnosed with a primary diagnosis of SCLC (extensive or limited) or stage III NSCLC, confirmed by pathology, between 1st of January 2015 and 31st of December 2019.

  4. Medical records available at the participating site reflect at least nine months of follow-up from the index date (unless the patient died within the first nine months of diagnosis)

Exclusion Criteria:

* 1. Patients with concomitant cancer at the time of diagnosis other than SCLC or stage III NSCLC, except for non-metastatic non-melanoma skin cancers, or in situ or benign neoplasms. Cancer will be considered concomitant if it occurs within five years of NSCLC or SCLC diagnosis 2. Patients initially diagnosed with stage I to II NSCLC who have progressed to stage III 3. Current or prior use of "Durvalumab" treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who were diagnosed with primary Small Cell Lung Cancer (Extensive stage & Limited Stage) or stage III Non-Small Cell Lung Cancer
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Treatment patterns of patients diagnosed with primary Small Cell Lung Cancer "SCLC" | 9 Month
  To characterize the treatment patterns of patients diagnosed with primary Small Cell Lung Cancer "SCLC" (Extensive stage & Limited Stage) through recoding type of treatment received
To characterize the treatment patterns of patients diagnosed with primary stage III Non-Small Cell Lung Cancer "NSCLC". | 9 Month
  To characterize the treatment patterns of patients diagnosed with primary stage III Non-Small Cell Lung Cancer "NSCLC". through recoding type of treatment received

SECONDARY OUTCOMES:
Patient demographic for the patients diagnosed with primary SCLC | 9 Months
  Recording Patient demographic for the patients diagnosed with primary SCLC (Age, gender, etc..)
Clinical characteristics for the patients diagnosed with primary SCLC | 9 Months
  Recording Clinical characteristics for the patients diagnosed with primary SCLC(Diagnosis, extent of the disease, etc...)
Patient demographic for patients diagnosed with primary stage III NSCLC | 9 Months
  Recording Patient demographic for patients diagnosed with primary stage III NSCLC(Age, gender, etc..)
Clinical characteristics for the patients diagnosed with primary stage III NSCLC | 9 Months
  Recording Clinical characteristics for the patients diagnosed with primary stage III NSCLC(Diagnosis, extent of the disease, etc...)

OTHER OUTCOMES:
Determining treatment effectiveness outcomes | 9 Months
  Determining treatment effectiveness outcomes:
  - Objective response rate [ORR]: is defined as the proportion of patients who have a partial or complete response to therapy; it does not include stable disease
Healthcare resource utilization (HCRU) associated with primary SCLC (Extensive stage & Limited Stage) / stage III NSCLC | 9 Months
  Recording healthcare resource utilization (HCRU) associated with primary SCLC (Extensive stage & Limited Stage) / stage III NSCLC treatment. HCRU will be assessed by describing the following:
  Hospitalizations, Outpatient visits, Emergency department visits, Number of medical and surgical treatments received, Use of imaging studies and other procedures
Determining treatment effectiveness outcomes | 9 Months
  Determining treatment effectiveness outcomes:
  - Disease control rate [DCR]: is a composite of ORR and stable disease

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4191R00036&attachmentIdentifier=f3baaaac-04b9-491c-a08a-b8f8c96fd013&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=